CLINICAL TRIAL: NCT01109134
Title: Prospective Randomized Controlled Clinical Study to Compare Tirofiban Intracoronary Bolus-Only vs Intravenous Bolus Plus Infusion in Patients With ST Elevation Myocardial Infarction Undergoing Primary Percutaneous Coronary Intervention
Brief Title: Tirofiban Intracoronary Bolus-only Versus Intravenous Bolus Plus Infusion in STEMI Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kosuyolu Heart Hospital (Other)
Collaborators: The Society of Cardiac Health Protection (Unknown)
Responsible Party: Cevat KIRMA, Kosuyolu Heart and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 33
Record Dates: First submitted 2010-04-21; First posted 2010-04-22 (Estimated); Last update posted 2010-04-22 (Estimated); Status verified 2010-03

CONDITIONS: Acute Myocardial Infarction
Keywords: primary angioplasty; tirofiban; microcirculation
MeSH Terms: interventions — Tirofiban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tirofiban intracoronary bolus-only (Experimental): Tirofiban bolus administered via intracoronary route at the time of primary PCI with no additional peri/postprocedural maintenance infusion
  Interventions: Drug: tirofiban intracoronary bolus-only
- Tirofiban intravenous bolus+infusion (Active Comparator): Tirofiban bolus administered intravenously before PCI, followed by periprocedural maintenance infusion
  Interventions: Drug: tirofiban intravenous bolus plus infusion

INTERVENTIONS:
Drug: tirofiban intracoronary bolus-only — administer tirofiban bolus intracoronary during primary percutaneous coronary intervention with no additional maintenance infusion
  Other Names: Aggrastat
  Arms: Tirofiban intracoronary bolus-only
Drug: tirofiban intravenous bolus plus infusion — administer tirofiban bolus intravenously and maintain infusion for up to 18 hours
  Other Names: Aggrastat
  Arms: Tirofiban intravenous bolus+infusion

SUMMARY:
The aim of this randomized trial is to compare the efficacy of high dose tirofiban administered as either an intracoronary bolus alone or as an intravenous bolus followed by a maintenance infusion with respect to microvascular perfusion and long term left ventricular infarct size, volumes and function.

DETAILED DESCRIPTION:
Primary percutaneous coronary intervention (PCI) is currently the treatment of choice for patients with acute ST elevation myocardial infarction (STEMI). Nevertheless, despite restoration of normal epicardial flow, myocardial perfusion remains impaired in approximately half of patients and is associated with a poor prognosis. A variety of invasive and non-invasive techniques have been proposed to evaluate microvascular perfusion and several invasive hemodynamic measures have been closely associated with microvascular damage.In order to improve microvascular perfusion after primary PCI, a variety of treatment strategies have been developed, such as adjunctive administration of glycoprotein IIb/IIIa inhibitors (GPIs). Although current ACC/AHA guidelines recommend that small molecule GPIs should be administered as a bolus followed by 18 hours of continuous infusion, changes in clinical practice may obviate the need for a maintenance infusion in current practice.

We hypothesized that when tirofiban is administered via intracoronary route, a bolus-only strategy may even be superior to intravenous bolus plus infusion strategy in maintaining myocardial perfusion. In order to evaluate microvascular function, we used a guidewire tipped with pressure and temperature sensors and measured the coronary hemodynamic parameters, as the index of microvascular resistance and coronary flow reserve, measures which have been closely associated with microvascular damage. In order to increase the predictive value of these indices, we performed these measurements four to five days after MI, because it has been shown that the extent of microvascular dysfunction changes, particularly within first 48 hours after reperfusion and stabilizes between 2 days and 1 week after perfusion

ELIGIBILITY:
Inclusion Criteria:

* Typical ongoing ischemic chest pain for longer than 30 minutes
* ST segment elevation of 0,1 mV or greater in at least two contiguous leads or a new left bundle branch block on the initial ECG.

Exclusion Criteria:

* Cardiogenic shock and / or clinical instability
* previous STEMI
* Malignant life threatening diseases
* Presence of an additional lesion causing more than 50% narrowing distal to the culprit lesion
* Contraindications to aspirin, clopidogrel, or heparin
* inability to give informed consent.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2008-09; Primary Completion 2009-02 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Indices of microvascular perfusion | Post-PCI day 4 to 5
  Intracoronary hemodynamic measures of index of microvascular resistance and coronary flow reserve

SECONDARY OUTCOMES:
ST segment resolution | post-PCI 90. minute
corrected TIMI frame count | immediately after PCI, post-PCI day 4 to 5
Myocardial Blush Grade | immediately after PCI, post-PCI day 4 to 5
Scintigraphic infarct size | 6th month
  Left ventricular infarct size by SPECT
Changes in left ventricular volume | Post-PCI day 3- 6th month
  Measured with echocardiography by using modified Simpson's method
Composite of major adverse cardiovascular events | 6 month
  composite of reinfarction, target vessel revascularization and death.

CONTACTS AND LOCATIONS:
Overall Officials: Cevat Kırma, Assoc.Prof, Study Chair — Kosuyolu Heart and Research Hospital; Ayhan Erkol, M.D, Principal Investigator — Kosuyolu Heart and Research Hospital